CLINICAL TRIAL: NCT00452257
Title: A Phase 1b Pharmacokinetic-Pharmacodynamic-Pharmacogenomic Study of Enzastaurin in Patients With B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: A Study of Enzastaurin in Patients With Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10724; H6Q-MC-S022
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Leukemia, Lymphocytic
MeSH Terms: conditions — Leukemia, Lymphoid | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: enzastaurin

INTERVENTIONS:
Drug: enzastaurin — 1125 mg loading dose then 500 mg, oral, daily, up to 3 years or until progressive disease
  Other Names: LY317615

SUMMARY:
The primary objective of this study is to see if enzastaurin affects the pGSK3 beta level in B-cell chronic lymphocytic leukemia (B-CLL) cells.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet all of the following criteria:

1. Patients with B-cell CLL as diagnosed by expression of CD19, CD5, and CD23 by flow cytometry.
2. Rai Stage III or IV disease or earlier stage disease with indications for therapy per NCI Working Group criteria (Cheson et al. 1996)
3. Absolute lymphocyte count > or = to 5,000/microliter, with a lymphocyte WBC differential of > or = to 70%.
4. Platelet count >20,000/microliter.
5. Adequate organ function, including the following:

   * Hepatic: bilirubin < or = to 1.5 times the upper limit of normal (x ULN); alkaline phosphatase (ALP), aspartate transaminase (AST), and alanine transaminase (ALT) < or = to 2.5 x ULN
   * Renal: serum creatinine < or = to 1.5 X ULN.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Are unable to swallow tablets.
2. Are unable to discontinue use of carbamazepine, phenobarbital, and phenytoin.
3. Are pregnant or breastfeeding.
4. Have central nervous system (CNS) metastases (unless the patient has completed successful local therapy for CNS metastases and has been off of corticosteroids for at least 4 weeks before starting study therapy).
5. Have a serious concomitant systemic disorder (including active bacterial, fungal, or viral infection) that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To characterize the inhibitory effects of enzastaurin on the pGSK3 beta level in B-CLL cells. | baseline, cycle 1, end of study

SECONDARY OUTCOMES:
Evaluation of activity of PKC beta in B-CLL cells | baseline, end of study
Response rate | baseline to measured progressive disease
Duration of response | time of response to progressive disease
Time to progressive disease | baseline to measured progressive disease
Safety | every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern Time (UTC/GMT- 5 hours,EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duarte, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com